CLINICAL TRIAL: NCT01996553
Title: The Prevalence of Radial Artery Occlusion in Diagnostic Cardiac Catheterization and Percutaneous Intervention
Status: Completed | Type: Observational
Sponsor: Jesse Brown VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Durham RN, BSN, CCRN, Registered Nurse, Jesse Brown VA Medical Center
Other Study IDs: 743024-6
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Coronary Angiography; Radial Artery Occlusion
Keywords: blood flow, regional; complications; disease, arterial obstructive; cardiac catheterization; radial artery
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transradial cardiac catheterization: Patients undergoing cardiac catheterization through the radial artery.

SUMMARY:
The purpose of this study is to establish the rate of radial artery occlusion post transradial cardiac catheterization through different modalities.

The study hypothesis is that specialized imaging can provide specific information to help identify hand complications after cardiac catheterization through the wrist.

DETAILED DESCRIPTION:
The purpose of this study is to establish the rate of radial artery occlusion post diagnostic/interventional cardiac catheterization through different modalities, and to compare current assessment methods (such as Allen's test, Modified Barbeau test and duplex ultrasonography) to specialized imaging techniques for sensitivity and specificity of radial artery occlusion detection post transradial catheterization.

The study hypothesis is that specialized imaging can provide a specific focused analysis of hand characteristics to identify physiologic abnormalities as a result of radial artery occlusion post transradial catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over the age of 18 who present to the Jesse Brown VA cath lab for a diagnostic radial artery angiogram or percutaneous intervention will be considered for the study.

Exclusion Criteria:

* Any subject who is unable to give informed consent or declines to participate will be excluded.
* Patients who have previously had a cardiac catheterization through the radial artery will be excluded because it will not be known if the changes to the circulation of the hand is secondary to the current or previous transradial catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects consist of patients who present to the cardiac catheterization laboratory for an angiogram or percutaneous intervention for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2013-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Physiologic abnormalities of the hand | 1 day to 3 weeks post transradial cardiac catheterization
  Blood flow to the hand in which transradial access was accomplished will be assessed for physiologic abnormalities as a result of radial artery occlusion post transradial catheterization
Physiologic abnormalities of the hand | 3 weeks to 3 months post transradial cardiac catheterization
  Blood flow to the hand in which transradial access was accomplished will be assessed for physiologic abnormalities as a result of radial artery occlusion

SECONDARY OUTCOMES:
Radial Artery Occlusion | 1 day to 3 weeks post transradial catheterization
  Radial artery blood flow will be assessed for patency or occlusion 1 day to 3 weeks post transradial cardiac catheterization
Radial Artery Occlusion | 3 weeks to 3 months post transradial catheterization
  Radial artery blood flow will be assessed for patency or occlusion 3 weeks to 3 months post transradial catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Durham, MS, APN, Principal Investigator — Jesse Brown VA Medical Center
Locations (1):
- Jesse Brown VA Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Barbeau GR, Arsenault F, Dugas L, Simard S, Lariviere MM. Evaluation of the ulnopalmar arterial arches with pulse oximetry and plethysmography: comparison with the Allen's test in 1010 patients. Am Heart J. 2004 Mar;147(3):489-93. doi: 10.1016/j.ahj.2003.10.038. PMID 14999199
- [Background] Durham KA. Cardiac catheterization through the radial artery. Am J Nurs. 2012 Jan;112(1):49-56. doi: 10.1097/01.NAJ.0000410370.81555.54. No abstract available. PMID 22222403
- [Background] Dandekar VK, Vidovich MI, Shroff AR. Complications of transradial catheterization. Cardiovasc Revasc Med. 2012 Jan-Feb;13(1):39-50. doi: 10.1016/j.carrev.2011.08.005. Epub 2011 Nov 23. PMID 22115936
- [Background] Sanmartin M, Gomez M, Rumoroso JR, Sadaba M, Martinez M, Baz JA, Iniguez A. Interruption of blood flow during compression and radial artery occlusion after transradial catheterization. Catheter Cardiovasc Interv. 2007 Aug 1;70(2):185-9. doi: 10.1002/ccd.21058. PMID 17203470
- [Background] Bazemore E, Mann JT 3rd. Problems and complications of the transradial approach for coronary interventions: a review. J Invasive Cardiol. 2005 Mar;17(3):156-9. No abstract available. PMID 15867445